CLINICAL TRIAL: NCT06368635
Title: The Cerebral Microcirculation Diseases and Coronary Microcirculation Disease Study（CCMD）
Brief Title: The Cerebral Microcirculation Diseases and Coronary Microcirculation Disease Study
Acronym: CCMD
Status: Recruiting | Type: Observational
Sponsor: Weijing Wang (Other Government)
Collaborators: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Sponsor-Investigator, Weijing Wang, Principal Investigator, China National Center for Cardiovascular Diseases
Organization: China National Center for Cardiovascular Diseases (Other Government)
Other Study IDs: 2022-GSP-QN-8
Record Dates: First submitted 2024-04-11; First posted 2024-04-16 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Microcirculation; Coronary Artery Disease; Cerebrovascular Circulation
MeSH Terms: conditions — Coronary Artery Disease | interventions — Coronary Angiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CCMD: The correlation between coronary microcirculation disease and cerebral microcirculation
  Interventions: Diagnostic Test: Coronary angiography

INTERVENTIONS:
Diagnostic Test: Coronary angiography — target vessel with intermediate coronary lesion (40-80% diameter stenosis and FFR(fractional flow reserve) ≥0.8； or severe stenosis（>80%）after successful PCI(percutaneous coronary intervention) and FFR ≥0.8

SUMMARY:
Ischaemic heart disease (IHD) and degenerative brain disease are two major sources of death and disability affecting all countries. While the consequences of obstructive disease in major vessels supplying blood to both organs have been widely documented, less attention has been paid to disease processes affecting the microcirculation that may affect cardiac and cerebral function. Yet, over the last decade significant progress has been made in understanding the substrate of microvascular disease in both organs. In the heart, arteriolar thickening and capillary rarefaction that reduce the conductance of the microvasculature and its ability to vasodilate in response to increased myocardial oxygen demands constitute the leading cause of coronary microvascular dysfunction (CMD). In the brain, concentric hyaline thickening of deep penetrating small arteries (arteriolosclerosis) with associated fibrosis of the vessel wall constitutes the most frequent substrate for cerebral small vessel disease (CSVD). Of note, both CMD and CSVD share common risk factors, such as age, hypertension, and diabetes.3 These factors might have a common effect on the microvascular domain of cardiac and cerebral vascular beds.

Although a potential link between both conditions has been hypothesized based on the similarities between pathological changes and risk factors, advance in knowledge exploring this has been hampered by lacking objective evidence of CMD and pathological brain changes indicative of CSVD in prior research studies. Thus, the relationship between CMD and CSVD is unknown.

The main objective of this study was to analyse the relationship between cerebrovascular disease and CMD in patients with atherosclerotic coronary artery disease (CAD).

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent available.
* Age 45-80 years.
* Stable coronary lesions.
* target vessel with intermediate coronary lesion (40-80% diameter stenosis and FFR ≥0.8； or severe stenosis（>80%）after successful PCI and FFR ≥0.8

Exclusion Criteria:

* Previous myocardial infarction in the territory of distribution of the target vessel.
* Aortic valve stenosis (moderate or severe) .
* Severe left ventricle hypertrophy.
* Left ventricle moderate systolic dysfunction (EF < 35%).
* Contraindications to adenosine.
* Previous CABG (Coronary artery bypass grafting) with permeable grafts.
* Contraindication to stent implantation.
* Severe anemia.
* Unilateral or bilateral carotid artery stenosis (> 50%).
* Unilateral or bilateral middle cerebral arteries (>50%).
* Previous cognitive decline, baseline MoCA less than 16 points.
* Coagulopathies or chronic anticoagulation.
* Platelets < 75000 o > 700.000.
* Previous stroke or intracranial hemorrhage.
* Contraindication to MRI.
* Chronic Renal Failure contraindicating gadolinium infusion during MRI: estimated glomerular filtration rate (eGFR) < 60 ml/min), hemodialysis, previous renal transplantation.
* Pacemaker/ Implantable Cardioverter Device with contraindication to MRI.
* Planned cardiac surgery.
* Life expectancy < 1 years.

Ages: 45 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with stable coronary lesions (stable coronary disease or lesions in nonculprit vessels >48 hours after acute coronary syndrome) with clinical indication to coronary angiography and intermediate coronary lesions (visual estimation) suitable for FFR-guided revascularization.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
MACE | 1 month
  Incidence of Major Cardiovascular Events (MACE): all-cause of death, myocardial infarction and any type of coronary revascularization
MACE | 12 month
  Incidence of Major Cardiovascular Events (MACE): all-cause of death, myocardial infarction and any type of coronary revascularization

SECONDARY OUTCOMES:
Cerebral microcirculation | baseline
  Determined by Cerebral MRI and Montreal Cognitive Assessment (MoCA) assessment. Montreal Cognitive Assessment (MoCA) The maximum score is 30 points, and the minimum score is 0 points. The lower the score, the more severe the cognitive impairment. A score of 26 or above is normal; 22-25 points: Mild cognitive decline; 16-21 points: Moderate cognitive decline; Below 16 points: Severe cognitive decline.
Cerebral microcirculation | 12 month
  Determined by Cerebral MRI and Montreal Cognitive Assessment (MoCA) assessment. Montreal Cognitive Assessment (MoCA) The maximum score is 30 points, and the minimum score is 0 points. The lower the score, the more severe the cognitive impairment. A score of 26 or above is normal; 22-25 points: Mild cognitive decline; 16-21 points: Moderate cognitive decline; Below 16 points: Severe cognitive decline.

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital, National Center for Cardiovascular Diseases, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
The person responsible for entering information about the study voluntarily provides these publications. These may be about anything related to the study.